CLINICAL TRIAL: NCT06158776
Title: Research on the Prediction and Mechanism of Rectal Adenoma Canceration Based on Radiomics of Multimodal MRI Combined With Clinical Indicators
Brief Title: Predicting Rectal Adenoma With Canceration and Investigating Mechanism Based on Multimodal MRI and Biochemical Model
Status: Completed | Type: Observational
Sponsor: Aiyin Li (Other)
Responsible Party: Sponsor-Investigator, Aiyin Li, professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: S1119
Record Dates: First submitted 2022-12-23; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Rectal Adenoma
Keywords: Rectal Adenoma;Canceration;Magnetic resonance imaging; Radiomics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this retrospective study is to establish a diagnostic model for rectal adenoma canceration. The model will include multimodal comprehensive HR-T2WI morphological score, IVIM functional imaging and radiomics features, and clinical indicators such as tumor markers, serum Gelsolin protein and peripheral blood inflammatory cell ratio. It can be to provide accurate diagnostic information for patients before surgery, which is of great value for formulating personalized treatment plans and improving the prognosis of patients.

DETAILED DESCRIPTION:
Imaging tests is the main method for evaluating rectal mass, especially MRI, which has been widely used in the preoperative diagnosis of rectal mass disease due to its very good soft tissue resolution. Previous studies in our group found that HR-T2WI-based radiomics, HR-T2WI-based morphology, and IVIM-based functional imaging can be used for the diagnosis of adenoma canceration. In addition to imaging, other tests, such as peripheral blood tests, can also reflect the development and progression of adenocarcinoma by counting tumor markers (colorectal tumor markers mainly CEA, AFP, CA199, CA724, CA50, CA242), inflammatory cell ratio (lymphocyte/C-reactive protein ratio, neutrophil/lymphocyte ratio, lymphocyte/monocytes ratio), and special types of proteins (such as coagulant protein).This study identifies the progression of adenoma to carcinoma by analyzing the combined cellular, morphological, and functional changes in adenoma carcinomas, with the expectation that multimodal co-diagnosis will improve the accuracy of clinical diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. surgical resection
2. pathologically confirmed rectal adenoma or rectal adenoma with canceration
3. rectal MRI examination including IVIM-DWI, within two weeks before surgery

Exclusion Criteria:

1. preoperative treatment
2. poor image quality, including intestinal gas or fecal artifact and IVIM image fitting error
3. no surgical resection but colonoscopy
4. pathologically confirmed rectal cancer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Collect patients who come to our hospital for surgery due to rectal mass, and preoperative colonoscopy is diagnosed as adenoma or suspected adenoma cancerous, and did not receive any treatment before surgery. Exclusion criteria: patients with malignant tumors of other organs, patients who have received neoadjuvant chemoradiotherapy before surgery, patients with other acute and chronic inflammation, and claustrophobia.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
morphological scoring based on HR-T2WI | 5-10 minutes
  Radiologists interpret the lesion according to the performance of HR-T2WI, and the interpretation criteria are whether the mucosal layer signal is continuous, whether the intestinal wall is wrinkled, and whether the tumor has external convexity.
IVIM parameter | 10-15 minutes
  IVIM sequence images were analyzed using Functool MADC software, and the region of interest (ROI) was placed in the solid region of the tumor, continuously outlining the edges of the hypertensive lesions. The D, D, and F values of the lesion are then measured and recorded.
Radiomics score | 10-15 minutes
  Tumor volume is manually sketched as ROI by RadCloudv2.2 platform on HR-T2WI images. Three sets of features were extracted based on VOI, and then the screened feature values were scored using software R.
Clinical indicators | 3-7 minutes
  The levels of tumor markers and inflammatory cell indexes of all patients in this study were collected, and meaningful indicators were statistically analyzed as one of the identification items. Tumor markers mainly include CEA, AFP, CA199, CA724, CA50 and CA242，inflammatory cell ratios include lymphocyte/C-reactive protein ratio, neutrophil/lymphocyte ratio and lymphocyte/monocytes ratio, in addition to special types of proteins (such as coagulant protein).

SECONDARY OUTCOMES:
Nomogram | 10-20 minutes
  Radiomics features were extracted based on tumor volume and screened to obtain meaningful features. Finally, the radiomics feature scores were obtained by weighted calculation as omics parameters.The T2 morphological score, IVIM parameters, meaningful clinical indicators and weighted omics scores were used as relevant factors to construct a concise nomogram for predicting the canceration of rectal adenoma.

CONTACTS AND LOCATIONS:
Overall Officials: Aiyin Li, Ph.D., Study Director — Qianfoshan Hospital
Locations (1):
- Qianfoshan Hosptial, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No